CLINICAL TRIAL: NCT04265950
Title: Multicenter, Randomized, Open-Label Trial in Children and Adolescents to Establish Optimal Number of Doses for HPV Vaccination in Children and Adolescents Living With HIV
Brief Title: Establishing Optimal Number of Doses for HPV Vaccination in Children and Adolescents Living With HIV, OPTIMO Trial
Acronym: OPTIMO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Asociación Civil Via Libre, Peru (Other); Evandro Chagas National Institute of Infectious Diseases (INI), Oswaldo Cruz Foundation (FIOCRUZ) (Unknown); National Cancer Institute (NCI) (NIH); GHESKIO Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RG1007065; U54CA242977 (NIH); NCI-2020-01098 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10521 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-02-07; First posted 2020-02-12 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: HIV Infection
Keywords: HPV vaccination; HIV infected children
MeSH Terms: conditions — HIV Infections | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Arm 1 (3 doses of 9vHPV vaccine) (Experimental): Participants living with HIV receive recombinant human papillomavirus nonavalent vaccine IM at enrollment, and at 2 and 6 months. Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 30 months.
  Interventions: Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm 2 (2 doses of 9vHPV vaccine) (Experimental): Participants living with HIV receive recombinant human papillomavirus nonavalent vaccine IM at enrollment and at 6 months. Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 30 months.
  Interventions: Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm 3 (1 dose of 9vHPV vaccine) (Experimental): Participants living with HIV receive recombinant human papillomavirus nonavalent vaccine IM at enrollment. Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 24 months and recombinant human papillomavirus nonavalent vaccine completion dose IM at 30 months.
  Interventions: Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm 4 (1 dose of 9vHPV vaccine) (Active Comparator): Participants without HIV receive recombinant human papillomavirus nonavalent vaccine IM at enrollment . Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 24 months and recombinant human papillomavirus nonavalent vaccine completion dose IM at 30 months.
  Interventions: Biological: Recombinant Human Papillomavirus Nonavalent Vaccine

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine

SUMMARY:
This phase IV trial compares 3 different dosing schedules to find the optimal number of doses for HPV vaccination in children and adolescents living with HIV. Comparing 3 different dosing schedules may help researchers determine whether a single dose of HPV vaccine could be effective in preventing HPV in children and adolescents living with HIV.

DETAILED DESCRIPTION:
OUTLINE: Participants living with HIV are randomized to one of three arms. HIV-negative participants are assigned to a fourth arm.

ARM 1: Participants living with HIV receive recombinant human papillomavirus nonavalent vaccine intramuscularly (IM) at enrollment, and at 2 and 6 months. Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 30 months.

ARM 2: Participants living with HIV receive recombinant human papillomavirus nonavalent vaccine IM at enrollment and at 6 months. Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 30 months.

ARM 3: Participants living with HIV receive recombinant human papillomavirus nonavalent vaccine IM at enrollment. Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 24 months and recombinant human papillomavirus nonavalent vaccine completion dose IM at 30 months.

ARM 4: Participants without HIV receive recombinant human papillomavirus nonavalent vaccine IM at enrollment. Participants also receive recombinant human papillomavirus nonavalent vaccine booster dose IM at 24 months and recombinant human papillomavirus nonavalent vaccine completion dose IM at 30 months.

ELIGIBILITY:
Inclusion Criteria:

* ARMS 1-3: Children must be living with HIV. HIV infection documented by positive molecular test or positive serologic test.
* ARM 4: Children must be healthy (e.g., without autoimmune disease or cancer) and not infected with HIV
* ARMS 1-3: Children must be on a consistent, clinically appropriate combination antiretroviral therapy (ART) regimen for > 6 months prior to study enrollment
* Children must be 9-13 years-old (at or after 9th birthday, prior to 14th birthday) at enrollment. This will allow vaccination of participants within the recommended age range for receipt of HPV vaccination in Peru and Brazil. Only children ages 9-11 (at or after 9th birthday, prior to 12th birthday) will be enrolled into arms 3 and 4
* Clinical laboratory values for children in Arms 1, 2, & 3 (CLWH) must be as described below:

  * CD4% >15% or CD4 counts >200 cells/ mm3
  * VL (<400 copies/mL)
* All female participants must not be pregnant (all females will receive pregnancy tests at all vaccine visits prior to receipt of study vaccine). The effects of Gardasil 9 on the developing human fetus at the recommended therapeutic dose are unknown. If pregnancy is confirmed during the screening process, enrollment will not occur. If pregnancy occurs after the first vaccine dose, additional vaccine doses will not be administered, but the child will remain in study follow-up.
* We anticipate that all children will enter the study prior to sexual debut. Sexual debut will be ascertained by participant questioning in Haiti. Physical examination will not be performed at any of the study sites. Potential participants who report sexual activity will not be enrolled
* Children in all arms must have the ability to understand and the willingness to assent to the study. Parents or guardians must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Children who have a serious illness requiring treatment with systemic medications other than ART (excluding short course oral steroids or inhaled steroid treatment for asthma), are currently under immunomodulatory therapy, received immunosuppressive therapy (> 10 mg/day of prednisone or equivalent for > 1 week) in the 6 months prior to enrollment date
* Children who received any vaccine within 3 weeks prior to enrollment date (these children will be encouraged to enroll after 3 weeks have passed)
* Children who received blood-derived products within 6 months prior to enrollment or planned use during the study period
* Children who weigh less than 18 kilograms
* Children with cancer being treated with chemotherapy or radiation
* Potential participants receiving any other investigational agents may be excluded in the opinion of the supervising physician
* Children in all arms with contraindications to vaccination, including pregnancy or breastfeeding
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Children having received HPV vaccination before study entry
* Children with evidence of sexually transmitted HIV infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to HPV vaccination

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Human papillomavirus type 16 (HPV16) neutralizing antibody geometric mean titers (GMTs) (Arm 1 versus [vs.] Arm 2) | At 24 months after the last dose of each vaccine regimen
  Pseudovirion (PsV)-based neutralization assays will be used to establish HPV 16 neutralizing antibody GMT.

SECONDARY OUTCOMES:
Human papillomavirus type 18 (HPV18) neutralizing antibody GMTs (Arm 1 vs. Arm 2) | At 24 months after the last dose of each vaccine regimen
  Pseudovirion (PsV)-based neutralization assays will be used to establish HPV 18 neutralizing antibody GMT.
Change in HPV16 and HPV18 binding antibody median fluorescence intensity-MFI (slope) (Arm 1 vs. Arm 2) | Between 1 month after the last dose and 18 months after the last dose, and between 18 months and 24 months after the last dose of each vaccine regimen
  The Luminex immunoassay-based assay will be used to measure HPV 16 and HPV 18 binding antibody MFI.
HPV16 and HPV18 neutralizing antibody GMTs (Arm 2 vs. Arm 3) | At 24 months after the last vaccine dose
  Pseudovirion (PsV)-based neutralization assays will be used to establish HPV 16 and HPV 18 neutralizing antibody GMT.
Change in HPV16 and HPV18 binding antibody MFI (slope) (Arm 2 vs. Arm 3) | Between 1 month and 18 months after the last vaccine dose, and between 18 months and 24 months after the last vaccine dose
  The Luminex immunoassay-based assay will be used to measure HPV 16 and HPV 18 binding antibody MFI.
Binding antibody MFI to all 9 vaccine HPV types (Arm 2 vs. Arm 3) | At month 7 in Arm 2 and month 25 in Arm 3
  Compare the response to a 0, 6- months two-dose schedule vs. a 0, 24-months two-dose schedule in children living with HIV (CLWH). The Luminex immunoassay-based assay will be used to measure HPV 16 and HPV 18 binding antibody MFI, as well as the binding antibody MFI for other HPV types.
HPV16 and HPV18 neutralizing antibody GMTs (Arm 3 vs. Arm 4) | At 24 months after the first (single) vaccine dose
  Pseudovirion (PsV)-based neutralization assays will be used to establish HPV 16 and HPV 18 neutralizing antibody GMT.
Change in HPV16 and HPV18 binding antibody MFI (slope) (Arm 3 vs. Arm 4) | Between 1 month and 18 months after the single vaccine dose, and between 18 months and 24 months after the first (single) vaccine dose
  The Luminex immunoassay-based assay will be used to measure HPV 16 and HPV 18 binding antibody MFI.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Duerr, MD, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- Evandro Chagas National Institute of Infectious Diseases (INI), Oswaldo Cruz Foundation (FIOCRUZ) STD and AIDS Clinical Research Laboratory, Rio de Janeiro, Rio de Janeiro, Brazil
- GHESKIO Center, Port-au-Prince, Haiti
- Via Libre, Lima, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinto-Santini D, Jalil EM, Fernandes GT, Hilaire G, Kolevic L, Cabello R, Grinsztejn B, Pape W, Deschamps MM, House MG, Brofsky E, Sahasrabuddhe VV, Dasgupta S, Pasalar S, Madeleine MM, Carter J, Prabhu PR, Galloway D, Duerr A. ULACNet-301, OPTIMO protocol: optimizing HPV vaccination regimen for cancer prevention in children and adolescents living with HIV. BMC Cancer. 2025 Jan 27;25(1):151. doi: 10.1186/s12885-025-13551-z. PMID 39871186

DOCUMENTS (1):
  • Informed Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT04265950/ICF_000.pdf